CLINICAL TRIAL: NCT07133061
Title: The Influence of Red Bull Energy Drink on the Speed, Strength and Rebound Performance of Female Volleyball Players at the Performance Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Bohemia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: USouthBohemiaKTVS
Record Dates: First submitted 2025-08-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Effect of Supplementation on Performance
Keywords: Volleyball; Energy drink; Wingate test; Jumping ergometry; Dynamometer; Comparison of the result

STUDY DESIGN:
Intervention Model Description: Each participant underwent both tests, with Redbull and with placewbo, in random order.
Who Masked: Participant
Masking Description: After enrollment in the study (in a pre-selected order of tests), participants were assigned a number under which they passed the tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Red Bull (Experimental): The group of participants performed a test after using Red Bull
  Interventions: Diagnostic Test: Wingate test; Diagnostic Test: Dynamometry; Diagnostic Test: Rebound plate; Diagnostic Test: Blood lactate test
- Without Red bull (Active Comparator): The group of participants performed a test after using a placebo
  Interventions: Diagnostic Test: Wingate test; Diagnostic Test: Dynamometry; Diagnostic Test: Rebound plate; Diagnostic Test: Blood lactate test

INTERVENTIONS:
Diagnostic Test: Wingate test — During the test, 1s power, 5s power, 30s power, speed, heart rate, the value of lactate and other parameters are determined.
Diagnostic Test: Dynamometry — The test determines the strength of the handshake by right and left hand separately.
Diagnostic Test: Rebound plate — The test determines the height of the jump from the right lower limb and from the left lower limb separately.
Diagnostic Test: Blood lactate test — Measurement of volume of lactate in the blood.

SUMMARY:
The first league female volleyball players of team VK Madeta České Budějovice were tested. Participants understood and agreed to the conditions of testing. The research group consisted of 15 female volleyball players aged 18-26 years,

DETAILED DESCRIPTION:
Participants The first league female volleyball players of team VK Madeta České Budějovice were tested. Participants understood and agreed to the conditions of testing. The research group consisted of 15 female volleyball players aged 18-26 years, who train 3 times a week and play matches almost every weekend, always on Fridays and Saturdays. All tested players completed all measurements and had no long breaks in the training process. According to the posts, 5 outside hitters, 4 blockers, 4 liberos and 2 setters. 3 players were left-handed and 12 were right-handed were tested. The average age was 21.3 ± 2.4 years, height 172.6 ± 5.8 cm, weight 70.2 ± 7.9 kg, BMI 23.6 ± 2.5 kg/m2, amount of fat 24.9 ± 5.6% and the amount of muscle mass 41.9 ± 3.2%. Somatic parameters from the first measurement were used to characterize the ensemble. The resulting values from the second measurement were identical and are therefore not included in the article. The participants underwent testing in the Laboratory of Load Diagnostics at Department of Sport Studies at the University of South Bohemia in the middle of the volleyball game season. Participants were healthy individuals with no known disability or injury and where in the full training process.

Ethical approval

The research was carried out with the consent of the Ethics Committee, Faculty of Education, University of South Bohemia, Ref. No.: 032//2023. All procedures performed in the study were in accordance with the ethical standards of the institutional research committee.

Measures, design and procedures

This is a retrospective study. The tested substance, namely a Red Bull brand energy drink and a placebo were provided during the testing. In the preparatory phase of the experiment, the placebo was prepared by mixing it on our own based on an inspiration from a similar testing in the USA, so that the taste and consistency of the drink resembled the Red Bull energy drink as much as possible. The recipe itself contained Schweppes Ginger Ale sparkling drink, granulated lemon tea and lemon-flavored beverage concentrate. The amount of both drinks served was determined individually depending on the weight of each of the tested players.

The determined weights of the players were averaged. The resulting average weight was 70 kg. After that, a simple mathematical calculation was used to find out the amount of fluid administered per kg of weight. The placebo contained Ginger Ale Schweppes in the same amount as Red Bull was administered and was further enriched with 20 g of lemon granulated tea and 5 ml of lemon concentrate. The drinks in opaque bottles with straws were served so that no difference was visually noticeable when serving the drink. The randomization tool GraphPad was used to divide the probands into two random groups. One group Red Bull was gave in the first round of testing and the other a placebo, and then reversed the process in the second round of testing.

The essential criterion for accurate testing was the individual's state of health and compliance with predetermined conditions. Participants were not supposed to eat for at least an hour before the test itself and should arrive after a good night's sleep. Each player was tested twice with a one-week break between measurements. The somatic parameters were measured first using the Inbody 770 device and the BSM 370 altimeter in underwear. After the somatic measurements, the player dressed in sports clothes in peace and gave her a pre-mixed drink to consume. She had about 3 minutes to drink it. After consuming the drink, the timer for 20 minutes was started and left the player in the resting phase. Participants waited for the caffeine to absorb into bloodstream. Once they consume an energy drink, it takes about 10 minutes for the caffeine to enter our bloodstream and their heart rate and blood pressure to rise. The time when caffeine levels peak in the bloodstream is 15-45 minutes. After 30-50 minutes, all the caffeine is fully absorbed. The same process with a caffeine-free placebo drink was applied. After the timer expired, there was a 5-minute warm-up in the sports hall, including a 2-minute-long run, 10 squats, 10 pull-ups and 1 minute of jumping rope in any way. After the warm-up, the testing was started. The first test was a manual dynamometry while sitting with a straight back. The KERN MAP dynamometer was used and tested the maximum grip of the right and left hand. The tested person always had two attempts for each hand. The measured values were noted in a pre-created table. After obtaining all the results, we always chose the better trial of the right and the left hand, after consuming the Red Bull energy drink and the placebo. The values of the right-hand press after consuming the Red Bull energy drink with the values after consuming a placebo were compared. The same for the left-hand pressure values was did.Next measurement was the Bosc test, which was performed in sports shoes on the Lode ProJump board. The participant standed on her right leg repeated the same, standing on her left leg and next on both of legs. After collecting all the results, the values after consuming the Red Bull drink were again compared with the values after consuming the placebo. The last measurement was the Wingate test on a bicycle ergometer LODE excalibur. First the POLAR chest belt was put on the player and adjusted the ergometer according to her physical parameters. The whole test was explained, including lactate sampling, so the participants knew all the instructions. The warm-up pedaling in the Wingate test lasted 5 min with a sustained pace of 60 rpm (revolutions per minute) and two, as fast as possible, climbs above 120 rpm. After 5 minutes, the main phase of the test followed. The participant reached maximum acceleration and tried to maintain it for 30 seconds. After that, the participant had 3 minutes of no-load ride with a maintaining pace of 60 rpm. Then we took blood lactate sample 30 seconds after the end of the test and asked the participant to rate the difficulty of the test according to Borg's method. The values of the lactate concentration were written down in a pre-prepared table, otherwise all data were forwarded to the computer. Using the Wingate test, the anaerobic parameters of individual players were determined. The resulting values, measured after drinking the Red Bull and the placebo were compared. The values of maximum heart rate, maximum relative power, average relative power, maximum 5s power, revolutions, fatigue index, lactate and evaluation according to the Borg scale were compared. At the end we asked the participants if they felt nauseous after drinking the beverage and noted the answer. Eight probands did not like the real Red Bull energy drink and they felt slightly nauseous after consuming it during testing. The entire measurement procedure in the same process, in order to obtain the most accurate results was repeated.

ELIGIBILITY:
Inclusion Criteria:

* age
* member of the team in the 1. league in volleyball
* female

Exclusion Criteria:

* acute illness

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is carried out on the female's volleyball team
Enrollment: 15 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Red Bull's influence on performance | Day 1 and day 8 (after 1 week, at the same time - second test).
  The aim of this study was to determine the acute effects of Red Bull energy drink consumption on speed, strength, rebound performance, anaerobic capacity, fatigue, physiological responses, and selected motor abilities in female volleyball players. Specifically, we evaluated its impact on performance and fatigue index in the Wingate anaerobic test, post-exercise blood lactate concentration, perceived exertion using the Borg scale, lower limb power assessed by Bosco's test, and maximal handgrip strength measured by hand dynamometry.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Bohemia, České Budějovice, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The data associated with the paper are not publicly available but are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once the article is published.
Access Criteria: If the article is in Open access mode, it will be accessible to all.